CLINICAL TRIAL: NCT06980467
Title: A Study on the Evaluation of Artificial Intelligence-Generated Clinical Advisory Outputs in Medical Professional Contexts
Brief Title: Evaluation of AI-Generated Clinical Advice by Physicians
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Tien Yin Wong, Vice-Provost and Senior Vice-Chancellor, Tsinghua University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2025-07
Record Dates: First submitted 2025-04-28; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Artificial Intelligence (AI)
MeSH Terms: interventions — Large Language Models

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Participants evaluate clinical recommendations generated by Language Model A (LLM-A), with subsequent assessments of communication style characteristics using rating scales.
- intervention group (Experimental): Participants evaluate clinical recommendations generated by Language Model B (LLM-B), followed by evaluations of communication style characteristics through metric instruments.
  Interventions: Other: Large Language Model

INTERVENTIONS:
Other: Large Language Model — An artificial intelligence system generating clinical recommendations using prompts, designed to simulate clinical advisory outputs. The protocol focuses on structured medical language generation.
  Arms: intervention group

SUMMARY:
This study examines how artificial intelligence systems interact with medical professionals. Researchers will compare physician responses to different AI-generated outputs in simulative medical scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Licensed physician or medical professional qualified to perform clinical evaluations;
* Willing to sign informed consent and commit time to participate in the study.

Exclusion Criteria:

* Unable to dedicate sufficient time to complete the study tasks;
* Unable or unwilling to understand and follow study instructions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-05-22 (Estimated); Study Completion 2025-05-23 (Estimated)

PRIMARY OUTCOMES:
Physician Response to AI-Generated Medical Content | Through study completion, an average of 1 week
  Participants will rate their level of agreement with AI-generated clinical suggestions presented in simulated medical scenarios. Responses will be recorded using a standardized rating scale (range 1-5, where higher scores indicate better agreement).

SECONDARY OUTCOMES:
Physician Perception of Communication Quality in AI-Generated Content | Through study completion, an average of 1 week
  Participants will assess the communication style of AI-generated content, focusing on factors such as empathy. Ratings will be collected using a standardized 5-point scale (range 1-5, where higher scores reflect higher perceived quality).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tsinghua University, Beijing, Beijing Municipality
  - Shanghai Health and Medical Center, Wuxi, Jiangsu